CLINICAL TRIAL: NCT05704673
Title: Effect of IV Nalbuphine on Postoperative Nausea and Vomiting Following Intrathecal Morphine in Patients Undergoing Inguinal Hernia Repair
Brief Title: Effect of IV Nalbuphine on Nausea and Vomiting Following Intrathecal Morphine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Marzouk Gomaa, house officer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17101956
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Inguinal Hernia
Keywords: nalbuphine; morphine; IV; Intrathecal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Longitudinal Studies; Double-Blind Method; Nalbuphine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Active Comparator): who given intrathecal morphine thin IV nalbuphine and asize of 80 patients
  Interventions: Drug: nalbuphine on N and V and pain with intrathecal morphine onInguinal hernia repair surgery. randomized, prospective, double blinded and placebo-controlled trial study.
- group (2) (Placebo Comparator): who given intrathecal morphine onInguinal hernia druing spinal anathesia
  Interventions: Drug: nalbuphine on N and V and pain with intrathecal morphine onInguinal hernia repair surgery. randomized, prospective, double blinded and placebo-controlled trial study.

INTERVENTIONS:
Drug: nalbuphine on N and V and pain with intrathecal morphine onInguinal hernia repair surgery. randomized, prospective, double blinded and placebo-controlled trial study. — investigate the effect of Iv nalbuphine on postoperative nausea and vomiting and pain with intrathecal morphine on inguinal hernia repair surgery.
  Other Names: nalbuphine; intrathecal morphine

SUMMARY:
the study aimed to investigate the effect of Iv nalbuphine on postoperative nausea and vomiting and pain with intrathecal morphine on inguinal hernia repair surgery.

DETAILED DESCRIPTION:
Bupivacaine hydrochloride is a commonly used local anesthetic in spinal anesthesia, however, the duration of spinal analgesia by bupivacaine is limited to about 75- 150 minutes.2 Therefore, various additives have been used with bupivacaine to prolong its effects and improve the quality of analgesia.(1) Opioids are the most popular used adjuvants added to bupivacaine in spinal blockade to obtain a sufficient intraoperative visceral analgesia and increase the duration and quality of postoperative analgesia, with less sympathetic block and hemodynamic effect .(2) morphine is commonly used for analgesia, but is frequently associated with postoperative nausea and vomiting (PONV) and pruritus, These side effects may lead to patient discomfort and prolonged hospital stay thus limiting the usefulness of IT morphine.

Nalbuphine is a mu receptor antagonist and a ĸappa receptor agonist.10 When added as an adjunct to intrathecal local anesthetics, it provides good analgesia with decreased incidence and severity of mu receptor side effects(3) Morphine binds most readily to the mu-opioid receptor and less well to the kappa-opioid receptor. So, the undesirable adverse events of morphine are thought to result from agonism at the mu-opioid receptor.5 Many drugs have been tried with morphine to potentiate its analgesic effects or to reduce the adverse events.6 Nalbuphine is a mixed opioid agonist-antagonist that acts mainly through kappa-opioid receptors, and it may attenuate mu-opioid receptor related side effects.3 Moreover, recent studies suggested that the analgesic effects of morphine and nalbuphine may be additive.

The addition of nalbuphine to intrathecal bupivacaine plus morphine significantly reduced the incidence and severity of postoperative nausea and vomiting and pruritus without affecting analgesic potency..(4)

ELIGIBILITY:
Inclusion Criteria:

* patients of aged 15-70years old
* males
* Scheduled patients for inguinal hernia repair surgery with under spinal anesthesia.
* ASA grade 1,2
* normal cardiac and renal function

Exclusion Criteria:

* Patient refusal
* Allergy to the studied drugs.
* Patients with contraindications to spinal anesthesia
* ASA grade 3,4

Ages: 15 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — males
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Effect of IV nalbuphine on postoperative nausea and vomiting following intrathecal morphine in patients undergoing inguinal hernia repair | 1. a. Primary (main): postoperative nausea and vomiting [ Time Frame: 24 hours ] A verbal descriptive scale (VDS) was used to assess the severity of PONV. ( no nausea=0, severe nausea= 3 by postoperative nausea and vomiting scale which range (o no nasuea
  investigate the effect of Iv nalbuphine on postoperative nausea and vomiting and pain with intrathecal morphine on inguinal hernia repair surgery.
  A verbal descriptive scale (VDS) was used to assess the severity of PONV. ( no nausea=0, severe nausea= 3 by postoperative nausea and vomiting scale which range (o no nasuea to 3 sever vomating).
  A verbal descriptive scale (VDS) was used to assess the severity of PONV b. Secondary (subsidiary): postoperative pain and puririts. [ Time Frame: 24 hours ] c. Visual analogue scale (VAS) pain scores (no pain = 0, worst possible pain = 3).

REFERENCES:
- [Result] Ibrahim AS, Aly MG, Thabet ME, Abdelaziz MR. Effect of adding nalbuphine to intrathecal bupivacaine with morphine on postoperative nausea and vomiting and pruritus after elective cesarean delivery: a randomized double blinded study. Minerva Anestesiol. 2019 Mar;85(3):255-262. doi: 10.23736/S0375-9393.18.12751-9. Epub 2018 May 30. PMID 29856176